CLINICAL TRIAL: NCT03495674
Title: CYCling Lynch Patients for Exercise and Prevention: CYCLE-P
Brief Title: Cycling in Preventing Colorectal Cancer in Participants With Lynch Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1035; NCI-2018-01046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-1035 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: High-Frequency Microsatellite Instability; Mismatch Repair Gene Mutation; Mutation-Negative Lynch Syndrome; Mutation-Positive Lynch Syndrome
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (FITBIT, cycling) (Experimental): Starting on day 15, participants wear FITBIT and complete cycling classes over 45 minutes 3 times a week for a total of 12 classes a month for up to 1 year.
  Interventions: Behavioral: Exercise Intervention; Device: Monitoring Device; Other: Questionnaire Administration
- Group II (FITBIT, information) (Active Comparator): Starting on day 15, participants receive information about exercise guidelines and wear FITBIT to track heart rate and activities for up to 1 year.
  Interventions: Other: Informational Intervention; Device: Monitoring Device; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Complete cycling classes
  Arms: Group I (FITBIT, cycling)
Other: Informational Intervention — Receive information about exercise guidelines
  Arms: Group II (FITBIT, information)
Device: Monitoring Device — Wear Fitbit
  Other Names: Monitor
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial studies how well cycling works in preventing colorectal cancer in participants with Lynch syndrome. Exercise such as cycling may reduce colorectal cancer risk in participants with Lynch syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of a 12-month exercise cycling intervention among Lynch syndrome (LS) patients.

SECONDARY OBJECTIVES:

I. To assess the effect size of exercise on circulating biomarkers as well as regulation of genomic, transcriptomic, and immunologic biomarkers in normal intestinal mucosa of LS patients.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Starting on day 15, participants wear FITBIT and complete cycling classes over 45 minutes 3 times a week for a total of 12 classes a month for up to 1 year.

GROUP II: Starting on day 15, participants receive information about exercise guidelines and wear FITBIT to track heart rate and activities for up to 1 year.

After completion of study interventions, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Lynch syndrome defined as meeting any of the following: (1) Mutation-positive Lynch syndrome: carriers or obligate carriers (by pedigree) of a pathogenic mutation in one of the deoxyribonucleic acid (DNA) mismatch repair (MMR) genes (i.e. MLH1, MSH2/EPCAM, MSH6, or PMS2) or (2) Mutation-negative Lynch syndrome: patients with a personal history of a non-sporadic MMR deficient premalignant lesion (i.e. polyp) or a non sporadic MMR deficient malignant tumor (where non-sporadic MMR deficient is defined by: microsatellite instability high by either immunohistochemistry or microsatellite instability (MSI) testing or both, but no evidence of MLH1 promoter methylation in cases with loss of both MLH1 and PMS2, and/or no evidence of BRAF mutation in cases with loss of both MLH1 and PMS2) but germline MMR genetic testing showed either a variant of unknown significance or mutation negative result or had declined germline MMR genetic testing.
* Participants must not have evidence of active/recurrent malignant disease for a minimum of 6 months.
* Participants must be at least 6 months from any prior cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy, hormonal therapy or radiation).
* Participants must have endoscopically accessible distal colon and/or rectal mucosa (i.e. participants must have at least part of the descending/sigmoid colon and/or rectum intact).
* Participants must consent to two standard of care lower gastro-intestinal GI endoscopy (flexible sigmoidoscopy or colonoscopy) with biopsies that will be 12 months (+/-21 days) apart.
* Ability to understand and the willingness to sign a written informed consent document.
* Must have normal cardiopulmonary exercise test prior to exercise participation.

Exclusion Criteria:

* Individuals who are status post total proctocolectomy (i.e. removal of all colon and rectum).
* Individuals with history of myocardial infarction, stroke, coronary-artery bypass draft, invasive coronary revascularization, arrhythmia requiring treatment such as atrial fibrillation, congestive heart failure, peripheral vascular disease, pulmonary embolism, or deep venous thrombosis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals with a history of diabetes, hypertension, or have smoked cigarettes in the last 12 months.
* Individuals who are unable to participate in cycling due to musculoskeletal limitations.
* Individuals who are unable to identify cycling classes in their community for exercise.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 1 year
  Defined as the proportion of eligible patients who consent to the number of patients who are contacted. This study will be considered as feasible if the recruitment rate is at least 20%.
Adherence rate | Up to 1 year
  Defined as the proportion of the actual attendance number to the planned number of exercise sessions (12 sessions monthly x 12 months) where patients will be required to comply with duration (time) of each session participated as well as monthly attendance. This study will be considered as feasible if the adherence rate is at least 75%.
Retention | Up to 1 year
  Defined as the proportion of participants who stay until study completion. This study will be considered as feasible if the retention rate is at least 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar-Sanchez, BLS,MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org